CLINICAL TRIAL: NCT06721156
Title: A Phase 2 Randomized, Placebo-Controlled, Double-Blind, Parallel-group Study to Evaluate the Efficacy and Safety of MK-1167 as Adjunctive Therapy in Participants With Mild to Moderate Alzheimer's Disease Dementia
Brief Title: A Study to Evaluate the Efficacy and Safety of MK-1167 in Participants With Alzheimer's Disease Dementia (MK-1167-008)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1167-008; 2024-515539-31-00 (Registry Identifier: EU CT); U1111-1309-3391 (Registry Identifier: UTN); jRCT2031240682 (Registry Identifier: jRCT)
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Alzheimer Disease; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MK-1167 3 mg (Experimental): Participants receive 3 mg of MK-1167 once daily (QD) for up to approximately 24 weeks.
  Interventions: Drug: MK-1167
- MK-1167 1 mg (Experimental): Participants receive 1 mg of MK-1167 QD for up to approximately 24 weeks.
  Interventions: Drug: MK-1167
- MK-1167 0.3 mg (Experimental): Participants take 0.3 mg of MK-1167 QD for up to approximately 24 weeks.
  Interventions: Drug: MK-1167
- Placebo (Placebo Comparator): Participants take placebo QD for up to approximately 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-1167 — MK-1167 oral capsule
  Arms: MK-1167 0.3 mg; MK-1167 1 mg; MK-1167 3 mg
Drug: Placebo — Placebo oral capsule
  Arms: Placebo

SUMMARY:
Researchers want to learn if giving MK-1167 (the study medicine) along with acetylcholinesterase inhibitor (AChEI) therapy can improve symptoms of Alzheimer's disease dementia (AD dementia), such as memory and mental activity. AD dementia is the most common type of dementia. AChEI therapy is the standard treatment for AD dementia.

The goals of this study are to learn:

* If at least one dose level (amount) of MK-1167 works to improve a person's memory and thinking compared to a placebo
* About the safety of MK-1167 and if people tolerate it

ELIGIBILITY:
Inclusion Criteria:

* Has mild to moderate Alzheimer's Disease (AD) dementia (ie, Stage 4 or Stage 5 AD) based on the Alzheimer's Association Revised Criteria for Diagnosis and Staging of Alzheimer's Disease
* Has a Mini-Mental State Examination (MMSE) score of 12 to 24 (inclusive)
* Is using acetylcholinesterase inhibitors (AChEI) therapy for management of AD dementia
* Has a designated study partner who can fulfill the requirements of this study. The study partner will need to spend sufficient time with the participant to be familiar with their overall function and behavior and be able to provide adequate information about the participant needed for the study including, knowledge of functional and basic activities of daily life, work/educational history, cognitive performance, emotional/psychological state, and general health status

Exclusion Criteria:

* Has a known history of stroke or cerebrovascular disease
* Has diagnosis of a clinically relevant central nervous system (CNS) disease other than AD dementia or other condition that negatively impacts cognition or cognitive status chronically
* Has structural brain disease
* Has a history of seizures or epilepsy
* Has any other major CNS trauma, or infections that affect brain function (eg, Human immunodeficiency virus (HIV), syphilis, and/or neurological sequelae of Coronavirus disease caused by severe acute respiratory syndrome coronavirus 2 (COVID-19), including impact on cognition)
* Has major medical illness or unstable medical condition
* Has a history of malignancy
* Resides in a nursing home or assisted care facility with need for direct continuous medical care and nursing supervision (with protocol-specified exceptions)
* Has liver disease, including but not limited to chronic viral hepatitis, nonviral hepatitis, cirrhosis, malignancies, autoimmune liver diseases

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in the Alzheimer's Disease Assessment Scale-11-item Cognitive Subscale (ADAS-Cog11) Total Score at Week 24 | Baseline and up to approximately 24 weeks
  The change from baseline in ADAS-Cog11 score at Week 24 is presented. ADAS-Cog11 is a structured scale that evaluates memory, orientation, attention, reasoning, language, and constructional praxis. ADAS-Cog11 measures cognition by assessing 11 metrics impaired in AD: word recall; commands; constructional praxis; naming objects and fingers; ideational praxis; orientation; word recognition; remembering test instructions; spoken language ability; word-finding difficulty; and comprehension of spoken language. The total possible score ranges from 0 to 70, with higher scores indicating greater cognitive impairment. Negative values indicate improvement relative to baseline, and vice versa.
Number of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately 28 weeks
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Intervention Due to an AE | Up to approximately 24 weeks
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study treatment due to an AE will be reported.

SECONDARY OUTCOMES:
Alzheimer's Disease Cooperative Study Clinical Global Impression of Change (ADCS-CGIC) Overall Score at Week 24 | Baseline and up to approximately 24 weeks
  The overall score in ADCS-CGIC at Week 24 is presented. The ADCS-CGIC is a clinician-rated measure of change in global severity from baseline, scored from 1 (marked improvement) to 7 (marked worsening), where 4 indicates no change. The assessment focuses on clinicians' observations of change in the participant's cognitive, functional, and behavioral performance since the beginning of the study.
Change From Baseline in The Alzheimer's Disease Cooperative Study Activities of Daily Living (ADCS-ADL) Total Score at Week 24 | Baseline and up to approximately 24 weeks
  The change from baseline in ADCS-ADL score at Week 24 is presented. The ADCS-ADL is an informant-based measure of the participant's functional ability in activities of daily living (ADLs). The ADCS-ADL assesses the competence of participants with AD dementia in basic and instrumental ADLs. The ADCS-ADL is a 23-item scale that includes 6 basic ADL items and 17 instrumental ADL items that provide a total score ranging from 0 to 78, with a lower score indicating greater severity.
Change From Baseline in the ADAS-Cog11 Total Score at Week 12 | Baseline and up to approximately 12 weeks
  The change from baseline in ADAS-Cog11 score at Week 12 is presented. ADAS-Cog11 is a structured scale that evaluates memory, orientation, attention, reasoning, language, and constructional praxis. ADAS-Cog11 measures cognition by assessing 11 metrics impaired in AD: word recall; commands; constructional praxis; naming objects and fingers; ideational praxis; orientation; word recognition; remembering test instructions; spoken language ability; word-finding difficulty; and comprehension of spoken language. The total possible score ranges from 0 to 70, with higher scores indicating greater cognitive impairment. Negative values indicate improvement relative to baseline, and vice versa.
ADCS-CGIC Overall Score at Week 12 | Baseline and up to approximately 12 weeks
  The overall score in ADCS-CGIC at Week 12 is presented. The ADCS-CGIC is a clinician-rated measure of change in global severity from baseline, scored from 1 (marked improvement) to 7 (marked worsening), where 4 indicates no change. The assessment focuses on clinicians' observations of change in the participant's cognitive, functional, and behavioral performance since the beginning of the study.
Change From Baseline in the ADCS-ADL Total Score at Week 12 | Baseline and up to approximately 12 weeks
  The change from baseline in ADCS-ADL score at Week 12 is presented. The ADCS-ADL is an informant-based measure of the participant's functional ability in activities of daily living (ADLs). The ADCS-ADL assesses the competence of participants with AD dementia in basic and instrumental ADLs. The ADCS-ADL is a 23-item scale that includes 6 basic ADL items and 17 instrumental ADL items that provide a total score ranging from 0 to 78, with a lower score indicating greater severity.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (72):
- United States (28):
  - Banner Alzheimer's Institute ( Site 0110), Phoenix, Arizona
  - Irvine Clinical Research ( Site 0104), Irvine, California
  - Anderson Clinical Research ( Site 0164), Redlands, California
  - California Neuroscience Research ( Site 0118), Sherman Oaks, California
  - JEM Research Institute / Headlands Research Network ( Site 0108), Atlantis, Florida
  - Brain Matters Research-Neurology ( Site 0150), Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida ( Site 0152), Fort Myers, Florida
  - Indago Research & Health Center, Inc ( Site 0128), Hialeah, Florida
  - K2 Medical Research THE VILLAGES ( Site 0166), Lady Lake, Florida
  - K2 Medical Research ( Site 0103), Maitland, Florida
  - Premier Clinical Research Institute ( Site 0114), Miami, Florida
  - Aqualane Clinical Research ( Site 0116), Naples, Florida
  - Headlands Research Orlando ( Site 0169), Orlando, Florida
  - Brain Matters Research ( Site 0151), Stuart, Florida
  - K2 Medical Research ( Site 0165), Tampa, Florida
  - Columbus Memory Center ( Site 0197), Columbus, Georgia
  - CenExel iResearch, LLC ( Site 0134), Savannah, Georgia
  - Tandem Clinical Research ( Site 0101), Marrero, Louisiana
  - Pharmasite Research, Inc. ( Site 0167), Baltimore, Maryland
  - Quest Research Institute ( Site 0173), Farmington Hills, Michigan
  - Velocity Clinical Research, Syracuse ( Site 0125), East Syracuse, New York
  - Mid Hudson Medical Research ( Site 0191), New Windsor, New York
  - Flourish Research - Charlotte ( Site 0106), Matthews, North Carolina
  - Velocity Clinical Research - Raleigh ( Site 0123), Raleigh, North Carolina
  - Summit Research Network ( Site 0111), Portland, Oregon
  - Kerwin Medical Center ( Site 0159), Dallas, Texas
  - Grayline Research Center ( Site 0105), Wichita Falls, Texas
  - Northwest Clinical Research Center ( Site 0102), Bellevue, Washington
- Argentina (5):
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 0207), Mar del Plata, Buenos Aires
  - IDIM - Instituto de Diagnóstico e Investigaciones Metabólicas ( Site 0204), Buenos Aires, Buenos Aires F.D.
  - Hospital Italiano de Buenos Aires ( Site 0209), Buenos Aires, Buenos Aires F.D.
  - Instituto Geriatrico Nuestra Señora de Las Nieves ( Site 0208), Buenos Aires, Buenos Aires F.D.
  - Instituto Kremer ( Site 0202), Córdoba
- Canada (3):
  - Okanagan Clinical Trials ( Site 0001), Kelowna, British Columbia
  - Ottawa Memory Clinic ( Site 0004), Ottawa, Ontario
  - Toronto Memory Program ( Site 0006), Toronto, Ontario
- Italy (5):
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico-UOSD Malattie Neurodegenerative ( Site 0903), Milan, Lombardy
  - Fondazione IRCCS San Gerardo dei Tintori ( Site 0902), Monza, Monza E Brianza
  - Centro S Giovanni Di Dio Fatebenefratelli ( Site 0904), Brescia
  - Ospedale San Raffaele. ( Site 0901), Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore ( Site 0905), Roma
- Japan (10):
  - Association of Healthcare Corporation Koukankai Koukan Clinic ( Site 1510), Kawasaki, Kanagawa
  - Kawasaki Saiwai Clinic ( Site 1501), Kawasaki, Kanagawa
  - Hatsuta Neurology Clinic ( Site 1507), Hirakata, Osaka
  - Nagomi Clinic ( Site 1506), Toyonaka, Osaka
  - Takesato Hospital ( Site 1522), Kasukabe, Saitama
  - Iwaki Clinic ( Site 1518), Anan, Tokushima
  - Enomoto Internal Medicine Clinic(Chofu) ( Site 1503), Chōfu, Tokyo
  - Nozomi Memory Clinic ( Site 1504), Mitaka, Tokyo
  - Tokyo Metropolitan Institute for Geriatrics and Gerontology ( Site 1515), tabashi City, Tokyo
  - Itsuki Hospital ( Site 1502), Tokushima
- Netherlands (3):
  - Brain Research Center Den Bosch B.V. ( Site 1002), 's-Hertogenbosch, North Brabant
  - Brain Research Center. ( Site 1001), Amsterdam, North Holland
  - Brain Research Center Zwolle ( Site 1003), Zwolle, Overijssel
- South Korea (4):
  - Inha University Hospital ( Site 1601), Incheon
  - Seoul National University Hospital ( Site 1604), Seoul
  - Hanyang University Seoul Hospital ( Site 1605), Seoul
  - Asan Medical Center ( Site 1603), Seoul
- Spain (7):
  - Centro de Atención Especializada Oroitu ( Site 1211), Algorta, Bizkaia
  - Hospital de la Santa Creu i Sant Pau ( Site 1204), Barcelona, Catalonia
  - Hospital Universitario 12 de Octubre ( Site 1208), Madrid, Madrid, Comunidad de
  - Hospital Universitari i Politecnic La Fe ( Site 1202), Valencia, Valencia
  - Fundació ACE ( Site 1206), Barcelona
  - Hospital Universitari Vall D Hebron ( Site 1203), Barcelona
  - Hospital Universitario Virgen de la Macarena ( Site 1210), Seville
- United Kingdom (7):
  - Brain Sciences Scotland Life Sciences-Aberdeen ( Site 1402), Aberdeen, Aberdeen City
  - Scottish Brain Sciences ( Site 1401), Edinburgh, Edinburgh, City of
  - Moorgreen Hospital ( Site 1409), Southampton, Hampshire
  - Remind UK ( Site 1404), Bath, Somerset
  - Re:Cognition Health - Birmingham ( Site 1406), Birmingham
  - Windsor Research Unit ( Site 1403), Cambridge
  - Campus for Ageing and Vitality ( Site 1408), Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com